CLINICAL TRIAL: NCT03939923
Title: Role of Sugammadex as Reversal Agent in Patients Extubated Immediately After Isolated Coronary Artery Bypass Grafting Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Matthew Ellison, Co-Director Cardiovascular Anesthesiology, Associate Professor, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1806161309
Record Dates: First submitted 2019-02-02; First posted 2019-05-07 (Actual); Results first posted 2023-12-22 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Surgery; Coronary Artery Disease
Keywords: Coronary Artery Bypass Grafting Surgery; Sugammadex
MeSH Terms: conditions — Coronary Artery Disease | interventions — Rocuronium; Neostigmine; Glycopyrrolate; Sugammadex

STUDY DESIGN:
Intervention Model Description: Group 1 (control) will receive reversal with neostigmine (0.04-0.07 mg/kg up to 5 mg maximal dosage) and glycopyrrolate (0.07-0.015 mg/kg up to 1mg maximal dosage).
  Group 2 (treatment) will receive reversal with sugammadex 2 mg/kg.
Who Masked: Care Provider
Masking Description: The nurses in the cardiac intensive care unit will be blinded to treatment allocation (Group 1 or 2).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neostigmine/Glycopyrrolate (Active Comparator): Group 1: Intubation with rocuronium at 1.0-1.2 mg/kg (vitals maintained within 20% of baseline). Subjects may be re-dosed with rocuronium at 0.1-0.4 mg/kg during the procedure to maintain 1-2 twitches on train of four (TOF) watch monitor reading recorded every 15 minutes. Group 1 (control) will receive reversal with neostigmine (0.04-0.07 mg/kg up to 5 mg maximal dosage) and glycopyrrolate (0.07-0.015mg/kg up to 1 mg maximal dosage).
  Interventions: Drug: Rocuronium; Drug: Neostigmine; Drug: Glycopyrrolate
- Sugammadex (Active Comparator): Group 2: Intubation with rocuronium at 1.0-1.2 mg/kg (vitals maintained within 20% of baseline). Subjects may be re-dosed with rocuronium at 0.1-0.4 mg/kg during the procedure to maintain 1-2 twitches on train of four (TOF) watch monitor reading recorded every 15 minutes. Group 2 (treatment) will receive reversal with Sugammadex (2mg/kg).
  Interventions: Drug: Rocuronium; Drug: Sugammadex

INTERVENTIONS:
Drug: Rocuronium — Intubation with Rocuronium 1.0-1.2 mg/kg (vitals maintained within 20% of baseline. Subjects may be re-dosed with rocuronium at 0.1-0.4 mg/kg during the procedure.
Drug: Neostigmine — Reversal with neostigmine (0.04-0.07 mg/kg up to 5 mg maximal dosage)
  Arms: Neostigmine/Glycopyrrolate
Drug: Glycopyrrolate — Reversal glycopyrrolate (0.07-0.015mg/kg up to 1 mg maximal dosage)
  Arms: Neostigmine/Glycopyrrolate
Drug: Sugammadex — Reversal with Sugammadex (2mg/kg)
  Arms: Sugammadex

SUMMARY:
The purpose of this study is to examine whether the use of Sugammadex will reduce time from reversal to extubation and improve other post extubation outcomes in Coronary artery bypass grafting patients. This study is a prospective, clinical interventional, randomized single blinded single-center design. The nurses in the cardiac intensive care unit will be blinded to treatment allocation (Group 1 or 2).

DETAILED DESCRIPTION:
Enhanced recovery pathways and early extubation of subjects undergoing cardiac procedures has now become mainstay, especially with the advent of minimally invasive procedures .

To facilitate optimal recovery after extubation; muscle strength is vital to prevent reintubation, improved deglutition and quicker transition to lower oxygen requirements, and better respiratory and cardiac hemodynamics. It also expedites de-escalation of acuity of care. Several studies have shown residual muscle weakness after full reversal with neostigmine and glycopyrrolate. Sugammadex is a direct reversal agent and can provide superior muscle strength, which optimizes respiratory function thereby preventing atelectasis, hypoxia and potentially avoiding reintubation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 70 years
* American Society of Anesthesiology physical status I-4
* Isolated coronary artery bypass graft surgery (CABG)
* Ability to give written informed consent

Exclusion Criteria:

* Any other surgical procedure concomitant to CABG surgery
* Known or suspected neuromuscular disease/pre-existing weakness
* Creatinine clearance less than 30 ml/min
* Bradycardia of less than 40 beats/min
* Pregnancy, breastfeeding women
* Known or suspected allergy to BRIDION® (sugammadex),neostigmine, or rocuronium
* Patients with contraindications towards sugammadex, neostigmine, or rocuronium
* Patients included in another trial within the last 30 days
* Patients with legal guardians or surrogate decision-making
* Female Patients who refuse to use non-hormonal contraceptive method or back-up method of contraception (such as condoms and spermicides) for the next 7 days if receiving sugammadex.
* Patients undergoing emergency surgery
* Patient refusal
* Patients with ejection fraction <30%
* Patients with restrictive and obstructive lung disease
* Patients with obstructive sleep apnea
* Patients with Body Mass Index greater than 40

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- WVU Medicine, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Badhwar V, Esper S, Brooks M, Mulukutla S, Hardison R, Mallios D, Chu D, Wei L, Subramaniam K. Extubating in the operating room after adult cardiac surgery safely improves outcomes and lowers costs. J Thorac Cardiovasc Surg. 2014 Dec;148(6):3101-9.e1. doi: 10.1016/j.jtcvs.2014.07.037. Epub 2014 Jul 31. PMID 25173117
- [Background] Subramaniam K, DeAndrade DS, Mandell DR, Althouse AD, Manmohan R, Esper SA, Varga JM, Badhwar V. Predictors of operating room extubation in adult cardiac surgery. J Thorac Cardiovasc Surg. 2017 Nov;154(5):1656-1665.e2. doi: 10.1016/j.jtcvs.2017.05.107. Epub 2017 Jun 13. PMID 28711332
- [Background] Murphy GS, Szokol JW, Avram MJ, Greenberg SB, Shear TD, Vender JS, Parikh KN, Patel SS, Patel A. Residual Neuromuscular Block in the Elderly: Incidence and Clinical Implications. Anesthesiology. 2015 Dec;123(6):1322-36. doi: 10.1097/ALN.0000000000000865. PMID 26448469
- [Background] Murphy GS, Kopman AF. "To Reverse or Not To Reverse?": The Answer Is Clear! Anesthesiology. 2016 Oct;125(4):611-4. doi: 10.1097/ALN.0000000000001280. No abstract available. PMID 27496655
- [Background] Herbstreit F, Zigrahn D, Ochterbeck C, Peters J, Eikermann M. Neostigmine/glycopyrrolate administered after recovery from neuromuscular block increases upper airway collapsibility by decreasing genioglossus muscle activity in response to negative pharyngeal pressure. Anesthesiology. 2010 Dec;113(6):1280-8. doi: 10.1097/ALN.0b013e3181f70f3d. PMID 20980910
- [Background] Boon M, Martini C, Broens S, van Rijnsoever E, van der Zwan T, Aarts L, Dahan A. Improved postoperative oxygenation after antagonism of moderate neuromuscular block with sugammadex versus neostigmine after extubation in 'blinded' conditions. Br J Anaesth. 2016 Sep;117(3):410-1. doi: 10.1093/bja/aew246. No abstract available. PMID 27543551
- [Background] Pongracz A, Szatmari S, Nemes R, Fulesdi B, Tassonyi E. Reversal of neuromuscular blockade with sugammadex at the reappearance of four twitches to train-of-four stimulation. Anesthesiology. 2013 Jul;119(1):36-42. doi: 10.1097/ALN.0b013e318297ce95. PMID 23665915
- [Background] Paton F, Paulden M, Chambers D, Heirs M, Duffy S, Hunter JM, Sculpher M, Woolacott N. Sugammadex compared with neostigmine/glycopyrrolate for routine reversal of neuromuscular block: a systematic review and economic evaluation. Br J Anaesth. 2010 Nov;105(5):558-67. doi: 10.1093/bja/aeq269. Epub 2010 Oct 8. PMID 20935005
- [Background] Park ES, Lim BG, Lee WJ, Lee IO. Sugammadex facilitates early recovery after surgery even in the absence of neuromuscular monitoring in patients undergoing laryngeal microsurgery: a single-center retrospective study. BMC Anesthesiol. 2016 Aug 2;16(1):48. doi: 10.1186/s12871-016-0221-2. PMID 27484887
- [Background] Chambers D, Paulden M, Paton F, Heirs M, Duffy S, Craig D, Hunter J, Wilson J, Sculpher M, Woolacott N. Sugammadex for the reversal of muscle relaxation in general anaesthesia: a systematic review and economic assessment. Health Technol Assess. 2010 Jul;14(39):1-211. doi: 10.3310/hta14390. PMID 20688009
- [Background] Chambers D, Paulden M, Paton F, Heirs M, Duffy S, Hunter JM, Sculpher M, Woolacott N. Sugammadex for reversal of neuromuscular block after rapid sequence intubation: a systematic review and economic assessment. Br J Anaesth. 2010 Nov;105(5):568-75. doi: 10.1093/bja/aeq270. Epub 2010 Oct 11. PMID 20937718
- [Derived] Ellison MB, Statler A, Grose B, Sloyer D, Hayanga H, Ellison PR, Funke C. Reversal of neuromuscular blockade after coronary artery bypass grafting: a randomized control trial. BMC Anesthesiol. 2025 Dec 23;25(1):612. doi: 10.1186/s12871-025-03456-6. PMID 41437213

RESULTS

PARTICIPANT FLOW:
Groups:
- Neostigmine/Glycopyrrolate: Group 1: Intubation with rocuronium at 1.0-1.2 mg/kg (vitals maintained within 20% of baseline). Subjects may be re-dosed with rocuronium at 0.1-0.4 mg/kg during the procedure to maintain 1-2 twitches on TOF watch monitor reading recorded every 15 minutes. Group 1 (control) will receive reversal with neostigmine (0.04-0.07 mg/kg up to 5 mg maximal dosage) and glycopyrrolate (0.07-0.015mg/kg up to 1 mg maximal dosage).
  Rocuronium: Intubation with Rocuronium 1.0-1.2 mg/kg (vitals maintained within 20% of baseline. Subjects may be re-dosed with rocuronium at 0.1-0.4 mg/kg during the procedure.
  Neostigmine: Reversal with neostigmine (0.04-0.07 mg/kg up to 5 mg maximal dosage)
  Glycopyrrolate: Reversal glycopyrrolate (0.07-0.015mg/kg up to 1 mg maximal dosage)
- Sugammadex: Group 2: Intubation with rocuronium at 1.0-1.2 mg/kg (vitals maintained within 20% of baseline). Subjects may be re-dosed with rocuronium at 0.1-0.4 mg/kg during the procedure to maintain 1-2 twitches on TOF watch monitor reading recorded every 15 minutes. Group 2 (treatment) will receive reversal with Sugammadex (2mg/kg).
  Rocuronium: Intubation with Rocuronium 1.0-1.2 mg/kg (vitals maintained within 20% of baseline. Subjects may be re-dosed with rocuronium at 0.1-0.4 mg/kg during the procedure.
  Sugammadex: Reversal with Sugammadex (2mg/kg)
Period: Overall Study
Arm/Group | Neostigmine/Glycopyrrolate | Sugammadex
Started | 42 | 42
Completed | 36 | 35
Not Completed | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Neostigmine/Glycopyrrolate | Sugammadex | Total
Number analyzed (Participants) | 36 | 35 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (8.36) | 62.1 (8.77) | 61.8 (8.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 25 | 25 | 50
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Time to Extubation
Description: Time to extubation: West Virginia University Hospitals use an electronic medical record (EMR) to chart "procedure stop." The definition for "time to extubation" is from the time the investigators chart "procedure stop" to the time of "extubation".
Time Frame: 0 minutes of study drug to 3 days after study drug administration
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Neostigmine/Glycopyrrolate | Sugammadex
Number analyzed (Participants) | 36 | 35
Minutes | 10.4 (5.9) | 6 (4.7)

2. Secondary Outcome: Heart Rate
Description: Heart rate post-reversal prior to extubation
Time Frame: 0 minutes to 2 hours after study drug administration
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Neostigmine/Glycopyrrolate | Sugammadex
Number analyzed (Participants) | 36 | 35
beats per minute | 81.5385 (13.6302) | 81.1622 (10.9735)

3. Secondary Outcome: Blood Pressure (First Measurement of Systolic Blood Pressure Post Reversal)
Description: Blood pressure; measure of systolic blood pressure of subject is obtained post-reversal prior to extubation of trachea
Time Frame: 0 minutes to 2 hours after study drug administration
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Neostigmine/Glycopyrrolate | Sugammadex
Number analyzed (Participants) | 36 | 35
mmHg | 105.6 (18.2067) | 112.1 (14.939)

4. Secondary Outcome: Tidal Volume
Description: Tidal volume post-reversal prior to extubation
Time Frame: between 30 minutes to 1 hour after extubation
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Neostigmine/Glycopyrrolate | Sugammadex
Number analyzed (Participants) | 36 | 35
Liters | 1.16 (0.5957) | 1.0975 (0.4977)

5. Secondary Outcome: Peak Flow Rate
Description: Peak flow rate - measured by peak flow meter post-extubation at 30-60 mins
Time Frame: 30-60 minutes post-extubation
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Neostigmine/Glycopyrrolate | Sugammadex
Number analyzed (Participants) | 36 | 35
L/min | 1.4609 (0.9968) | 1.416 (0.8466)

6. Secondary Outcome: Swallowing Capacity
Description: In the intensive care unit: If the patient awake and alert, is able to be positioned, can cough when asked, able to follow command to lick top and bottom lip, and is able to breathe freely then a registered nurse bedside swallowing/dysphagia screen is performed at a time point somewhere between 30 and 60 minutes following the operating room extubation. To perform the screen, a teaspoon is used to place distilled water on each subject's tongue, 3 mL each time 2 consecutive times. Then 3 ounces of water intake. The patient is asked to swallow the water to evaluate the swallowing ability. Aspiration of fluid (choking) subjectively divided into 4 categories: normal, no choking or hoarse voice after swallowing; mild, no choking but slight hoarseness of voice; moderate, no choking but a clearly identifiable hoarseness of voice; severe, choking.
Time Frame: Between 30 and 60 minutes post-extubation
Measure: Count of Participants; unit: Participants
Arm/Group | Neostigmine/Glycopyrrolate | Sugammadex
Number analyzed (Participants) | 36 | 35
Participants
  Passed | 29 | 33
  No Pass | 4 | 2
  Not assessed | 3 | 0

7. Other Pre Specified Outcome: Oxygen Saturation
Description: Oxygen saturation post-extubation
Time Frame: 30 minutes post-extubation
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Post-extubation Oxygen Requirements
Description: Post-extubation Oxygen requirements in subsequent 2 hours
Time Frame: 2 hours post-extubation
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Length of Stay Cardiac Intensive Care Unit
Description: Length of stay in the cardiac intensive care from onset of reversal drugs
Time Frame: 0 days after study drug to 100 days after study drug
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Reintubation Incidence
Description: Reintubation incidence in the first 24 hours post-extubation
Time Frame: 24 hours post-extubation
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Occurrence of Postoperative Respiratory Complications
Description: Postoperative respiratory complication including re-intubation
Time Frame: 0 hours after study drug to 24 hours after study drug
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Occurrence of Postoperative Cardiac Complications
Description: Postoperative cardiac complications including myocardial infarction, arrythmias
Time Frame: from 0 hours after study drug to 2 hours after study drug
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected for a 24 hour period. The 24 hour period begins when surgery stop is designated in the electronic medical record.
Description: Defined as any unfavorable and unintended medical occurrence, symptom, or disease temporally associated with the use of a medical treatment of the subjects whether it is associated or related to the medical treatment. The Principal Investigator will identify and make adverse events assessments. Adverse events and severe adverse events such as pneumonia, arrhythmia, and reintubation within 24 hours will be compared in both groups.
Arm/Group | Neostigmine/Glycopyrrolate | Sugammadex
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/35
Serious Adverse Events (participants affected / at risk) | 2/36 | 1/35
Other Adverse Events (participants affected / at risk) | 1/36 | 1/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neostigmine/Glycopyrrolate (N=36) | Sugammadex (N=35)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0) — ST Segment Elevation (on EKG) Myocardial Infarction unrelated to study
R ICA Stroke (Vascular disorders) | 1 (1) | 0 (0) — Right Internal Carotid Artery Cerebrovascular Stroke unrelated to study
R MCA Stroke (Vascular disorders) | 0 (0) | 1 (1) — Right Middle Cerebral Artery Cerebrovascular Stroke unrelated to study
OTHER ADVERSE EVENTS (reported when occurring in more than 2.8% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neostigmine/Glycopyrrolate (N=36) | Sugammadex (N=35)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1) — Atrial Fibrillation not related to study
Incomplete Right Bundle Branch Block (Cardiac disorders) | 1 (1) | 0 (0) — Incomplete Right Bundle Brach Block not related to study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-09-25): https://cdn.clinicaltrials.gov/large-docs/23/NCT03939923/Prot_SAP_ICF_000.pdf